CLINICAL TRIAL: NCT05431738
Title: Esophageal Stent With or Without Anti-migration Device for Tumors of the Gastroesophageal Junction: Multicenter Randomized Controlled Study. ANTIMIG Study
Brief Title: Anti-Migration System for Anti-reflux Oeso-gastric Stent (ANTIMIG)
Acronym: ANTIMIG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société Française d'Endoscopie Digestive (Other)
Responsible Party: Principal Investigator, KARSENTI, Principal Investigator, Société Française d'Endoscopie Digestive
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANTIMIG
Record Dates: First submitted 2022-06-19; First posted 2022-06-24 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Stent Migration; GastroEsophageal Cancer
Keywords: Stent Migration; GastroEsophageal Cancer; Esophageal Stenosis; Esophageal cancer; Endoscopy
MeSH Terms: conditions — Esophageal Stenosis; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, controlled, randomized, multicentre, single-blind study.
Who Masked: Participant
Masking Description: The stent is placed under endoscopy during general anesthesia. The type of stent is not specified in the endoscopy report. The patient is not informed of the type of esophageal stent placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STENT WITH ANTI-MIGRATION DEVICE (Active Comparator): Placement of a gastroesophageal stent with anti-migration device : Ella®, Leufen, Novatech
  Interventions: Device: Gastroesophageal stent placement
- STENT WITHOUT ANTI-MIGRATION DEVICE (Active Comparator): Placement of a gastroesophageal stent without anti-migration device : Hanarostent® ECW, Life Partners Europe
  Interventions: Device: Gastroesophageal stent placement

INTERVENTIONS:
Device: Gastroesophageal stent placement — A gastroesophageal stent is placed during a digestive endoscopy performed under general anesthesia, under endoscopic and fluoroscopic control

SUMMARY:
The aim of this prospective, controlled, randomized, multicentre, single-blind study is to compare the rate of intragastric migration of 2 types of esophageal stents with and without an anti-migration device placed for locally advanced or metastatic malignant stenosis of the gastroesophageal junction.

DETAILED DESCRIPTION:
In order to reduce the rate of spontaneous intragastric migration of esophageal stent placed for gastroesophageal junction tumor, anti-migration device has been developed. Pilot studies suggest the absence of morbidity of this device, but no comparative study has been conducted to confirm the interest of this anti-migration device.

The aim of this study is to compare the rate of intragastric migration of 2 types of esophageal stents with and without an anti-migration device placed for locally advanced or metastatic malignant stenosis of the gastroesophageal junction.

* Main objective: To evaluate the rate of intragastric migration of 2 types of esophageal stents (one with and the second without anti-migration device) placed for malignant stenosis of the gastroesophageal junction.
* Secondary objective(s):

  * Degraded migration rate (M3 and M6) if patient alive, and duration of survival without dysphagia
  * Comparison of the morbidity of these two stents
  * Comparison of the effectiveness of these two stents on dysphagia and reflux
  * Clinical and technical failure rate of these two stents

This is a prospective, controlled, randomized, multicentre, single-blind study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient of both sexes aged 18 or over.
2. Patient admitted to one of the investigation centers for dysphagia due to tumoral stenosis of the gastroesophageal junction, locally advanced or metastatic.
3. Patient ASA 1, ASA 2, ASA 3
4. Absence of participation in another clinical study
5. Signed Informed Consent
6. Patients benefiting from the social security system.

Exclusion Criteria:

1. Patient referred for stenosis by extrinsic compression by an extra digestive mass
2. Patients with contraindications relating to the procedures essential for the introduction of a stent
3. Mediastinal radiotherapy or esophageal surgery history
4. Patient under 18 or over 90
5. Patient ASA 4, ASA 5
6. Pregnant Woman
7. Patient unable to give personal consent
8. Absence of signed informed consent

Ages: 18 Years to 91 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Stent Intragastric migration rate at M1 | 1 month
  Stent Intragastric migration rate at M1 confirmed on radiography or CT

SECONDARY OUTCOMES:
Stent Intragastric migration rate at M3 | 3 months
  Stent Intragastric migration rate at M3 confirmed on radiography or CT
Stent Intragastric migration rate at M6 | 6 months
  Stent Intragastric migration rate at M6 confirmed on radiography or CT
Dysphagia recurrence at M1 | 1 month
  Dysphagia evaluation in 5 stages (Atkinson score) at M1 0 - no dysphagia
  1. - Clinging to the swallowing of solids
  2. - Semi-liquid feeding possible
  3. - Liquid feeding possible
  4. - Aphagia (need for parenteral nutrition)
Dysphagia recurrence at M3 | 3 months
  Dysphagia evaluation in 5 stages (Atkinson score) at M3 0 - no dysphagia
  1. - Clinging to the swallowing of solids
  2. - Semi-liquid feeding possible
  3. - Liquid feeding possible
  4. - Aphagia (need for parenteral nutrition)
Dysphagia recurrence at M6 | 6 months
  Dysphagia evaluation in 5 stages (Atkinson score) at M6 0 - no dysphagia
  1. - Clinging to the swallowing of solids
  2. - Semi-liquid feeding possible
  3. - Liquid feeding possible
  4. - Aphagia (need for parenteral nutrition)
Dysphagia-free survival time | 3 years
  Dysphagia-free survival time at the end of the study
Technical success rate of stent placement | 1 day
  Technical success rate of stent placement under digestive endoscopy defined by good progression of contrast through the stent into the gastric cavity after stent placement
Clinical success rate of stent placement on dysphagia | 3 days
  Medical success rate of stent placement under digestive endoscopy on dysphagia (dysphagia resorption after endoscopy)
Gastroesophageal reflux disease (GERD) after stent placement | 1 month
  Gastroesophageal reflux disease with the Reflux Disease Questionnaire (RDQ) score. The Reflux Disease Questionnaire a 12-item self-administered questionnaire, was designed to assess the frequency and severity of heartburn, regurgitation, and dyspeptic complaints and to facilitate the diagnosis of GERD. Minimum 12 : better outcome Maximum 72 : worse outcome
Stent placement complication : hemorrhage | 7 days
  Necessity of blood transfusion and/or endoscopic management
Stent placement complication : pain | 7 days
  Need for opioid treatment for more than 48 hours after stent placement or removal of the stent because of pain
Stent placement complication : pneumoperitoneum | 1 day
  Pneumoperitoneum diagnosed by CT in case of abnormal pain within hours of stent placement

CONTACTS AND LOCATIONS:
Locations (1):
- French Society of Digestive Endoscopy, Paris, France